CLINICAL TRIAL: NCT03549637
Title: Prevalence of fAmilial hypobetalipopRoTeinemIa in psychiaTrIc pOpulatioN
Brief Title: Prevalence of fAmilial hypobetalipopRoTeinemIa in psychiaTrIc pOpulatioN (PARTITION)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC17_0468
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Familial Hypobetalipoproteinemia
Keywords: Psychiatry, hypobetalipoproteinemia, LDL-Cholesterol
MeSH Terms: conditions — Hypobetalipoproteinemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychiatric population (Experimental): At inclusion: Patients will have A Lipid Panel Test, other biological analyzes and a clinical assessment. In case of a low LDL-C level (≤ 0, 50 g/L), genetic analyzes will be performed to screen for genetic forms of hypobetalipoproteinemia (HBL).
  At 2- 4 weeks: for patients with HBL (LDL-C ≤ 0,50 g/L with no secondary cause of LDL-C reduction), another Lipid Panel Test will be performed to confirm the maintenance of the low LDL-C level.
  At 6 months : Patients with a HBL will perform a full biological examination, and the LDL-C levels and genetic analyzes will be confirmed. A dietary survey will be performed, together with a psychiatric assessment. The same numbers of matched controls will performed a quick telephone interview to collect the psychiatric characteristics.
  Interventions: Diagnostic Test: Psychiatric population

INTERVENTIONS:
Diagnostic Test: Psychiatric population — Genetic and biological analysis of patients

SUMMARY:
The links between low LDL-C levels and psychologic symptoms (psychotic disorders, mood disorders, aggressivity, suicidal risk, etc.) and cognitive deficits (mainly executing functioning) are debated. The PARTITION study aims at estimating the prevalence of hypobetalipoproteinemia (HBL), defined as a LDL-C level ≤ 0,50 g/L, in a psychiatric population.

DETAILED DESCRIPTION:
Some forms of hypobetalipoproteinemia (HBL) are associated with a longevity syndrome and cardiovascular protection due to prolonged exposure to low levels of LDL-C. However, while LDL-C reduction has been studied extensively for its beneficial effect on cardiovascular risk, other studies have reported that low levels of LDL-C (either spontaneous or artificially occurring with low-fat diets or lipid-lowering drugs) may be associated with psychiatric symptoms (psychotic or mood disorders, aggression, suicidal attempts, etc.) or altered cognitive performance (particularly executive functioning). These studies have led to contradictory results, and the possible link between low LDL-C levels and psychiatric symptoms remains highly controversial so far.

The PARTITION study aims at estimating the prevalence of hypobetalipoproteinemia (HBL), defined as a LDL-C level ≤ 0,50 g/L, in a psychiatric population. Moreover, the study includes the characterization of psychiatric disorders as well as psychological and personal characteristics associated with HBL. The evolutionary profile of patients with and without HBL will be studied. Genetic characteristics and biomarkers of HBL will also be studied.

ELIGIBILITY:
Inclusion Criteria:

All patients hospitalized in one of the full-time adult psychiatric departments of Nantes University Hospital may be included, without maximum age limit.

Minors and patients under guardianship and tutorship may be included, taking into account the study population and the low risks and constraints of the study

Exclusion Criteria:

* minors under 15 years
* pregnant or nursing woman;
* simultaneous participation in another interventional research on a drug;
* not mastering the reading and writing of the French language well enough

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of primary hypobetalipoproteinemia prevalence defined by a spontaneously low level of LDL-C | at baseline (admission at the hospital)
  LDL-C level < 0,50 g/L

CONTACTS AND LOCATIONS:
Overall Officials: Marie GRALL-BRONNEC, Pr, Principal Investigator — Nantes University Hospital Nantes
Locations (1):
- Nantes University Hospital Nantes, Nantes, France